CLINICAL TRIAL: NCT02229318
Title: A Taste and Acceptance Study of FruitiVits, for Use in the Dietary Management of Young Children Requiring Very Restrictive Diets Such as the Ketogenic Diet.
Brief Title: A Taste and Acceptance Study of FruitiVits in Children Aged 4-8 Years Following a Ketogenic Diet.
Acronym: FruitiVits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitaflo International, Ltd (Industry)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NA-FRV-012014-01
Record Dates: First submitted 2014-08-26; First posted 2014-09-01 (Estimated); Results first posted 2016-10-07 (Estimated); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: Seizure Disorders
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FruitiVits (Experimental): Daily administration of FruitiVits dietary supplement
  Interventions: Dietary Supplement: FruitiVits

INTERVENTIONS:
Dietary Supplement: FruitiVits — Daily administration of FruitiVits dietary supplement

SUMMARY:
Subjects will be asked to substitute their usual vitamin and mineral supplement/s with FruitiVits for seven consecutive days.

DETAILED DESCRIPTION:
The study will involve 12 subjects between 4 and 8 years of age, who routinely use comprehensive micronutrient supplementation as part of their dietary management.

Primary Hypothesis:

FruitiVits is an acceptable source of vitamin, mineral and trace elements for patients on a Ketogenic diet.

Secondary Hypothesis:

FruitiVits will be well accepted and tolerated when given orally to children on a Ketogenic diet.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of condition requiring a Ketogenic diet
2. Currently on a Ketogenic diet
3. Aged 4 - 8 years
4. Routinely taking a complete micronutrient supplement
5. Oral feeding

Exclusion Criteria:

1) Children aged less than 4 years or older than 9 years of age

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2014-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Bergqvist, M.D, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Division of Neurology, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children between the ages of 4 and 8 years, attending the Ketogenic Diet Center at The Children's Hospital of Philadelphia were invited by email to attend a study family day held on a Saturday afternoon in September 2014. The first 12 families to respond were contacted via telephone and invited to enroll in the study.
Pre-assignment Details: 12 families invited to participate, one subject failed to attend the recruitment family day and did not enroll in the study.
Period: Overall Study
Arm/Group | FruitiVits
Started | 11 (September 6th 2014 11 enrolled)
Completed | 11 (September 15th 2014 11 completed)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FruitiVits
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 6.7 [4.3 to 8.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of FruitiVits
Description: The study product was rated on a scale of 1-5:
  1. (liked very much)
  2. (liked moderately)
  3. (neither liked nor disliked)
  4. (disliked moderately)
  5. (disliked very much).
Time Frame: Day 8 of trial
Population: Children aged 4 to 8 years.
Measure: Number; unit: participants
Arm/Group | FruitiVits
Number analyzed (Participants) | 11
participants
  Appearance score 1-3 | 8
  Smell score 1-3 | 10
  Taste score 1-3 | 6
  Texture score 1-3 | 6

2. Secondary Outcome: Ease of Preparation of FruitiVits
Description: Ease of preparation of FruitiVits was rated on a scale of 1-5:
  1. (very easy)
  2. (moderately easy)
  3. (neither easy nor difficult)
  4. (moderately difficult)
  5. (very difficult).
  Those who considered it not difficult to prepare and scored 1-3 on the scale: 11/11 patients
Time Frame: Day 8 of trial
Population: Children aged 4 to 8 years.
Measure: Number; unit: participants
Groups:
- FruitiVits: Administration of FruitiVits dietary supplement
Arm/Group | FruitiVits
Number analyzed (Participants) | 11
participants | 11

ADVERSE EVENTS:
Time Frame: 7 days per patient
Description: A symptom diary was completed for each patient specifically asking about the following:
  Nausea and/or vomiting Diarrhea and/or constipation Gas, flatulence and/or regurgitation Abdominal bloating and/or distention Abdominal discomfort and/or pain
Arm/Group | FruitiVits
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No